CLINICAL TRIAL: NCT02772692
Title: Influence of Defecation Postures on Functional Consumption in Humans
Brief Title: Defecation Postures for Functional Consumption
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhanwei Zhao, Director, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20160511
Record Dates: First submitted 2016-05-11; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Squatting pan (Experimental): Defecation using a squatting pan
  Interventions: Behavioral: Squatting pan
- Toilet (No Intervention): defecation using a standard-sized toilet

INTERVENTIONS:
Behavioral: Squatting pan — Using squatting pans to replace standard-sized toilets in one group of the included constipation patients
  Arms: Squatting pan

SUMMARY:
Whether functional consumption is influenced by defecation postures is unclear. The investigators investigated effects of defecation postures on functional consumption.

DETAILED DESCRIPTION:
Constipation is a chronic problem in many patients all over the world. In some groups of patients such as the elderly, constipation is a significant health care problem. A prospective study was performed at 3 hospitals in China. The included patients were functional consumption patients with defecation sitting on a standard-sized toilet. Patients received standard functional consumption treatment according to the guideline and were randomly assigned to groups that using a squatting pan or a standard-sized toilet.

ELIGIBILITY:
Inclusion Criteria:

* Subject has functional constipation
* Subject does not receive other treatments

Exclusion Criteria:

* History of heart cerebrovascular disease
* History of other types of constipation
* Pregnant, trying to become pregnant or breast feeding
* Age< 18-year and >70-year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of defecation | Six months
  Frequency of defecation per week is collected by an interview questionnaire.

SECONDARY OUTCOMES:
Frequency of re-defecation after the first defecation | Six months
  Frequency of re-defecation after the first defecation per week is collected by an interview questionnaire.
Defecation time | Six months
  Defecation time (minute) is assessed by watch and collected by an interview questionnaire.
Sensation of non-complete defecation | Six months
  Sensation of non-complete defecation is investigated by an interview questionnaire (0: no; 1: yes).
Straining forces during defecation | Six months
  Straining forces during defecation is assessed by the rating of defecation exertion (0-1-2-3: very easy, easy, difficult, very difficult).

CONTACTS AND LOCATIONS:
Overall Officials: Qingchuan Zhao, MD, Principal Investigator — Xijing Hospital

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Roberts MC, Millikan RC, Galanko JA, Martin C, Sandler RS. Constipation, laxative use, and colon cancer in a North Carolina population. Am J Gastroenterol. 2003 Apr;98(4):857-64. doi: 10.1111/j.1572-0241.2003.07386.x. PMID 12738468
- [Result] Lindberg G, Hamid SS, Malfertheiner P, Thomsen OO, Fernandez LB, Garisch J, Thomson A, Goh KL, Tandon R, Fedail S, Wong BC, Khan AG, Krabshuis JH, LeMair A; World Gastroenterology Organisation. World Gastroenterology Organisation global guideline: Constipation--a global perspective. J Clin Gastroenterol. 2011 Jul;45(6):483-7. doi: 10.1097/MCG.0b013e31820fb914. No abstract available. PMID 21666546
- [Result] Rao SS, Kavlock R, Rao S. Influence of body position and stool characteristics on defecation in humans. Am J Gastroenterol. 2006 Dec;101(12):2790-6. doi: 10.1111/j.1572-0241.2006.00827.x. Epub 2006 Oct 6. PMID 17026568